CLINICAL TRIAL: NCT02951884
Title: The Effect of Intra-articular Local Anesthetic Injection and Hematoma Aspiration on Pain and Narcotic Analgesia Use Following Tibial Plateau Fractures
Brief Title: Intra-articular Local Anesthetic Injection and Hematoma Aspiration
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was stopped for feasibility (low enrollment)
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, William Lack, Assistant Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 208755
Record Dates: First submitted 2016-10-28; First posted 2016-11-01 (Estimated); Results first posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Tibial Fractures
Keywords: Aspiration; Bupivacaine; Epinephrine; Marcaine; Pain; Shin Bone
MeSH Terms: conditions — Tibial Fractures; Pain | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive aspiration of the joint alone, receive aspiration of the knee joint and an injection of 20cc bupivacaine 0.5% with 1:200,000 epinephrine, or receive no injection or aspiration therapy
Who Masked: Participant
Masking Description: This study uses a single blind masking scheme
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Aspiration (Experimental): Participants assigned to this arm receive aspiration of the joint alone in which a needle will be introduced into the knee joint to withdraw the blood that collects within the knee.
  Interventions: Procedure: Aspiration
- Aspiration with injection (Experimental): Participants assigned to this arm receive aspiration of the knee joint and an injection of 20cc bupivacaine 0.5% with 1:200,000 epinephrine
  Interventions: Procedure: Aspiration; Drug: Bupivacaine
- Control (No Intervention): Participants assigned to this arm receive no injection or aspiration therapy.

INTERVENTIONS:
Procedure: Aspiration — A needle is placed into the knee joint and all of the blood that is in the joint is removed.
  Arms: Aspiration; Aspiration with injection
Drug: Bupivacaine — An injection of 20cc bupivacaine 0.5% with 1:200,00 epinephrine
  Other Names: Marcaine; Exparel; Sensorcaine
  Arms: Aspiration with injection

SUMMARY:
The primary objective of this study is to determine whether a patient with a tibial plateau fracture (non-displaced, displaced, or depression type) will have decreased pain and narcotic analgesia requirements following an intra-articular injection of local anesthetic and aspiration of the knee.

DETAILED DESCRIPTION:
We propose to study tibial plateau fractures treated at our institution for which we have fracture data, treated with open reduction internal fixation (ORIF) procedures or treated non-operatively. Patients will be identified based on the classification of their injury, that being tibial plateau fracture; we will seek to sub-classify each patient based on the Shatzker classification of tibial plateau fractures and using knee osteoarthritis (OA) classification as our prospective study will be based on both tibial plateau fractures as a whole and their sub-classification: Lateral tibial plateau fracture without depression (I), lateral tibial plateau fracture with depression (II), compression fracture of the lateral (IIIA) or central (IIIB) tibial plateau, medial tibial plateau fracture (IV), bicondylar tibial plateau fracture (V), and tibial plateau fracture with diaphyseal discontinuity (VI). It is important for our prospective study to classify each fracture pattern as they generally differ in energy of injury and thus may affect pain management or need for narcotic pain medications and also potentially affect functional outcomes.

Following consent for participation in the study, patients will be blinded to initial management of the tibial plateau fracture with either: Aspiration of the joint alone, aspiration of the knee joint and injection of 20cc bupivacaine 0.5% with 1:200,000 epinephrine, or no injection or aspiration therapy for a control arm. Using the block randomization list, the patient will be randomized at the time of consent for participation. For the sake of consistency, all participating treating physicians (orthopaedic on-call residents) will be trained on Sawbones Fully Encased Knee Joint with Patella and Ligaments for a standardized aspiration and injection technique.

For the patients randomized into the treatment arms, the knee will be held in 15-30 degrees short of full extension and fully prepped using chlorhexidine wipes in a centrifugal manner. An 18 gauge spinal needle will be introduced into the superolateral aspect of the knee (if the knee is too edematous, an inferolateral or inferomedial approach may be appropriate). We will aspirate the knee with a 60cc syringe until we are unable to draw out more fluid and record the volume on a case record form. Subsequently, we will remove the syringe from the needle connection, leaving the 18 gauge needle in place. Then we will draw up 30cc of 0.5% bupivacaine with 1:200,000 epinephrine (Marcaine) with .18-gauge needle into the second 60cc syringe. Subsequently, we will place the filled syringe on the 18 gauge needle already in the knee and inject. Then we will remove the needle-syringe construct and place a bandage over the injection site.

The patient's initial numerical rating scale (NRS) score will be recorded immediately. Subsequent visual analogue scale (VAS) scores will be recorded at 5 minutes after intervention and at hours 2, 4, 6, 8, 12, and 24 after initial work-up of the patient. Patients treated as an outpatient will record these values themselves. Patients will be directed to bring the completed form with them to their regular clinic follow-up visit. Additionally, supplemental analgesia requirements will be recorded upon administration and will be converted to morphine equivalent units for analysis. All patients admitted to the orthopedic service will be placed on patient-controlled analgesic (PCA) morphine, where the dose is determined by the weight of the patient. All other patients (those admitted to other services) will have analgesia converted to Opioid Morphine Equivalents (OMEs).

ELIGIBILITY:
Inclusion Criteria:

* Patients with isolated tibial plateau fractures aged 18 years and older
* Patients with tibial plateau fractures and associated soft tissue complaints about the knee, not associated with a fracture outside of the tibial plateau
* Patients with bilateral tibial plateau fractures and no other noted fractures

Exclusion Criteria:

* Any patient that does not wish to participate in the study or is unable to give consent at the initial encounter
* Patients under 18 years old
* Pregnant patients
* Patients who are unable to understand the study procedures
* Incarcerated patients
* History of allergic reaction to local anesthetics
* Emergent conditions requiring operations or airway protection
* Polytrauma patients
* Patients presenting for care greater than 24 hours following their injury.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Lack, MD, Principal Investigator — Loyola University Chicago
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers

REFERENCES:
- [Background] Manidakis N, Dosani A, Dimitriou R, Stengel D, Matthews S, Giannoudis P. Tibial plateau fractures: functional outcome and incidence of osteoarthritis in 125 cases. Int Orthop. 2010 Apr;34(4):565-70. doi: 10.1007/s00264-009-0790-5. Epub 2009 May 14. No abstract available. PMID 19440710
- [Background] Koval KJ, Helfet DL. Tibial Plateau Fractures: Evaluation and Treatment. J Am Acad Orthop Surg. 1995 Mar;3(2):86-94. doi: 10.5435/00124635-199503000-00004. PMID 10790657
- [Background] Stein C, Comisel K, Haimerl E, Yassouridis A, Lehrberger K, Herz A, Peter K. Analgesic effect of intraarticular morphine after arthroscopic knee surgery. N Engl J Med. 1991 Oct 17;325(16):1123-6. doi: 10.1056/NEJM199110173251602. PMID 1653901
- [Background] Busch CA, Shore BJ, Bhandari R, Ganapathy S, MacDonald SJ, Bourne RB, Rorabeck CH, McCalden RW. Efficacy of periarticular multimodal drug injection in total knee arthroplasty. A randomized trial. J Bone Joint Surg Am. 2006 May;88(5):959-63. doi: 10.2106/JBJS.E.00344. PMID 16651569
- [Background] Franceschi F, Rizzello G, Cataldo R, Denaro V. Comparison of morphine and ropivacaine following knee arthroscopy. Arthroscopy. 2001 May;17(5):477-80. doi: 10.1053/jars.2001.19684. PMID 11337713
- [Background] Jaureguito JW, Wilcox JF, Cohn SJ, Thisted RA, Reider B. A comparison of intraarticular morphine and bupivacaine for pain control after outpatient knee arthroscopy. A prospective, randomized, double-blinded study. Am J Sports Med. 1995 May-Jun;23(3):350-3. doi: 10.1177/036354659502300318. PMID 7661266
- [Background] White BJ, Walsh M, Egol KA, Tejwani NC. Intra-articular block compared with conscious sedation for closed reduction of ankle fracture-dislocations. A prospective randomized trial. J Bone Joint Surg Am. 2008 Apr;90(4):731-4. doi: 10.2106/JBJS.G.00733. PMID 18381308
- [Background] Perdreau A, Joudet T. Efficacy of multimodal analgesia injection combined with corticosteroids after arthroscopic rotator cuff repair. Orthop Traumatol Surg Res. 2015 Dec;101(8 Suppl):S337-45. doi: 10.1016/j.otsr.2015.09.006. Epub 2015 Nov 10. PMID 26563923
- [Background] Chalidis BE, Papadopoulos PP, Sachinis NC, Dimitriou CG. Aspiration alone versus aspiration and bupivacaine injection in the treatment of undisplaced radial head fractures: a prospective randomized study. J Shoulder Elbow Surg. 2009 Sep-Oct;18(5):676-9. doi: 10.1016/j.jse.2009.04.003. Epub 2009 May 31. PMID 19487135
- [Background] Ditsios KT, Stavridis SI, Christodoulou AG. The effect of haematoma aspiration on intra-articular pressure and pain relief following Mason I radial head fractures. Injury. 2011 Apr;42(4):362-5. doi: 10.1016/j.injury.2010.09.003. Epub 2010 Oct 8. PMID 20932520
- [Background] Bijur PE, Latimer CT, Gallagher EJ. Validation of a verbally administered numerical rating scale of acute pain for use in the emergency department. Acad Emerg Med. 2003 Apr;10(4):390-2. doi: 10.1111/j.1553-2712.2003.tb01355.x. PMID 12670856
- [Background] Heard SO, Edwards WT, Ferrari D, Hanna D, Wong PD, Liland A, Willock MM. Analgesic effect of intraarticular bupivacaine or morphine after arthroscopic knee surgery: a randomized, prospective, double-blind study. Anesth Analg. 1992 Jun;74(6):822-6. doi: 10.1213/00000539-199206000-00008. PMID 1595914
- [Background] Badner NH, Bourne RB, Rorabeck CH, MacDonald SJ, Doyle JA. Intra-articular injection of bupivacaine in knee-replacement operations. Results of use for analgesia and for preemptive blockade. J Bone Joint Surg Am. 1996 May;78(5):734-8. doi: 10.2106/00004623-199605000-00013. PMID 8642030

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from June 2016 through May 2018 (24 months) from the Orthopaedic Surgery and Rehabilitation Center at Loyola University Medical Center.
Period: Overall Study
Arm/Group | Aspiration | Aspiration With Injection | Control
Started | 0 | 1 | 1
Completed | 0 | 1 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population comprises both participants who consented to participate in the trial
Groups:
- Total: Total of all reporting groups
Arm/Group | Aspiration | Aspiration With Injection | Control | Total
Number analyzed (Participants) | 0 | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0 | 0
  Between 18 and 65 years |  | 1 | 0 | 1
  >=65 years |  | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 0 | 0 | 0
  Male |  | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 | 0 | 0
  Not Hispanic or Latino |  | 1 | 1 | 2
  Unknown or Not Reported |  | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0 | 0
  Asian |  | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0 | 0
  Black or African American |  | 0 | 0 | 0
  White |  | 1 | 1 | 2
  More than one race |  | 0 | 0 | 0
  Unknown or Not Reported |  | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Numerical Rating Scale (NRS) Pain Scores
Description: Twenty-four hours after injury, patients will self report their numerical rating scale (NRS) score. The NRS score ranges from 0 to 10 with higher scores indicating greater pain.
Time Frame: 24 hours
Population: The analysis population comprises both participants who consented to participate in the trial
Measure: Number; unit: units on a scale
Arm/Group | Aspiration | Aspiration With Injection | Control
Number analyzed (Participants) | 0 | 1 | 1
units on a scale |  | 7 | 2

2. Secondary Outcome: Supplemental Analgesia
Description: Twenty-four hours after injury, the researchers will record the number of participants that required supplemental analgesia.
Time Frame: 24 hours
Population: The analysis population comprises both participants who consented to participate in the trial
Measure: Count of Participants; unit: Participants
Arm/Group | Aspiration | Aspiration With Injection | Control
Number analyzed (Participants) | 0 | 1 | 1
Participants | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from June 2016 through May 2018 (i.e., 24 months)
Description: Because no individuals were assigned to the aspiration group, no individuals in that group were at risk for adverse events or all cause mortality
Arm/Group | Aspiration | Aspiration With Injection | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
The study was stopped for feasibility (low enrollment)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-03): https://cdn.clinicaltrials.gov/large-docs/84/NCT02951884/Prot_SAP_000.pdf